CLINICAL TRIAL: NCT04797910
Title: Effect of Antiviral Therapy on HVPG in Patients With Viral Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2021-002
Record Dates: First submitted 2021-03-07; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Complications associated with portal hypertension are the leading cause of death in patients with cirrhosis. Until now, hepatic venous pressure gradient (HVPG) - the difference between the wedged hepatic venous pressure (WHVP) and the free hepatic vein pressure (FHVP)- has been the criterion standard to determine portal pressure. Antiviral therapy may decrease HVPG which needs to be verified.

ELIGIBILITY:
Inclusion Criteria:

* Patients with viral cirrhosis were diagnosed;
* Age 18-80 years;
* Need and willing to accept measure HVPG;
* First HVPG measurement of more than 5 mmHg;
* Signed Informed Consent

Exclusion Criteria:

* Patients with viral cirrhosis have been treated with antiviral therapy and have achieved virological response;
* Ready to accept or have accepted a TIPS procedure;
* Splenic embolization was performed;
* Inaccurate measurement of HVPG due to combined hepatic venous shunt;
* Complicated with alcoholic liver disease, autoimmune liver disease or other types of liver disease;
* Complicated with liver cancer or other organ malignancy;
* Combined with severe cardiopulmonary disease affects survival;
* Complicated with severe renal insufficiency;
* Concomitant portal vein cavernous degeneration or extensive portal vein thrombosis;
* Women who are planning to become pregnant or who are pregnant or breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatitis B cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-03-10 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
HVPG changed and reached the response standard | one year
  HVPG response to therapy indicates a decrease in HVPG of at least 10% from baseline or to less than 12 mmHg after chronic treatment with NSBBs.

SECONDARY OUTCOMES:
Antiviral therapy achieved a virological response | one year
  HBV-DNA remained undetectable for successive two times.

IPD SHARING:
Plan to Share IPD: No